CLINICAL TRIAL: NCT01363583
Title: Prostacyclin Treatment in Severe Traumatic Brain Injury: a Microdialysis and Outcome Study
Brief Title: Study on the Effect of Prostacyclin Compared to Placebo in Traumatic Brain Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Professor Lars-Owe Koskine, Umea university
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 151:633=01
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2001-09

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Epoprostenol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- epoprostenol, Flolan® (Active Comparator): Measurement on the effect of epoprostenol on lactate/pyruvate ratio measured by cerebral microdialysis
  Interventions: Drug: epoprostenol versus normal saline
- normal saline (Placebo Comparator): Effect of saline on the lactate/pyruvate ratio measured by cerebral microdialysis
  Interventions: Drug: epoprostenol versus normal saline; Drug: normal saline

INTERVENTIONS:
Drug: epoprostenol versus normal saline — 0.5 ng/kilogram/minute during 4 days
  Other Names: Flolan®; Normal saline
Drug: normal saline — 0.5-1.5 ml/hour during 4 days
  Arms: normal saline

SUMMARY:
This study is a prospective consecutive double-blinded randomized study on the effect of PGI2, prostacyclin (epoprostenol, Flolan®) versus placebo (saline)in patients with severe traumatic brain injury. All patients with severe traumatic brain injury were eligible for inclusion. Inclusion criteria: verified traumatic brain injury, Glasgow Coma Score (GCS) at intubation and sedation of ≤ 8, age 15-70 years, a first-recorded cerebral perfusion pressure (CPP) of > 10 mm Hg, and arrival within 24 hours after trauma.

Tne primary aim was to evaluate whether treatment with epoprostenol would reduce a lactate/pyruvate ratio,as measured by cerebral microdialysis after 24 hours of treatment.

A secondary aim was to evaluate the effect of epoprostenol on systemic inflammatory markers, measured by different cytokines.

ELIGIBILITY:
Inclusion Criteria:

* traumatic brain injury, Glasgow coma scale ≤ 8

Exclusion Criteria:

* pregnant or lactating women

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Lactate/pyruvate ratio 24 hours after start of epoprostenol versus placebo | 24 hours

SECONDARY OUTCOMES:
Levels of systemic inflammatory markers | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Owe Koskinen, Professor, Principal Investigator — Umea university
Locations (1):
- Umea university, Umeå, Sweden

REFERENCES:
- [Result] Olivecrona M, Rodling-Wahlstrom M, Naredi S, Koskinen LO. Prostacyclin treatment in severe traumatic brain injury: a microdialysis and outcome study. J Neurotrauma. 2009 Aug;26(8):1251-62. doi: 10.1089/neu.2008.0605. PMID 19226191
- [Derived] Hagglund L, Olivecrona M, Koskinen LD. Correlation of Cerebral and Subcutaneous Glycerol in Severe Traumatic Brain Injury and Association with Tissue Damage. Neurocrit Care. 2022 Jun;36(3):993-1001. doi: 10.1007/s12028-021-01412-z. Epub 2021 Dec 16. PMID 34914037
- [Derived] Olivecrona Z, Bobinski L, Koskinen LO. Association of ICP, CPP, CT findings and S-100B and NSE in severe traumatic head injury. Prognostic value of the biomarkers. Brain Inj. 2015;29(4):446-54. doi: 10.3109/02699052.2014.989403. Epub 2014 Dec 18. PMID 25518864
- [Derived] Wahlstrom MR, Olivecrona M, Ahlm C, Bengtsson A, Koskinen LO, Naredi S, Hultin M. Effects of prostacyclin on the early inflammatory response in patients with traumatic brain injury-a randomised clinical study. Springerplus. 2014 Feb 18;3:98. doi: 10.1186/2193-1801-3-98. eCollection 2014. PMID 24600548